CLINICAL TRIAL: NCT03582644
Title: Cryotherapy Effectiveness on Pain, Physical Function and Quality of Life in Individuals With End Stage Knee Osteoarthritis - a Case Series
Brief Title: Cryotherapy Effectiveness in Individuals With End Stage Knee Osteoarthritis - a Case Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Lucas Ogura Dantas, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 81166517.7.0000.5504
Record Dates: First submitted 2018-06-26; First posted 2018-07-11 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; Cryotherapy; Physiotherapy; Physical Agent
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Cryotherapy; Ice

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRYOTHERAPY INTERVENTION (Experimental): Patients with end stage knee osteoarthritis, both sexes, 60 years or higher
  Interventions: Other: Cryotherapy

INTERVENTIONS:
Other: Cryotherapy — Crushed ice (1kg) inside a plastic bag (24x34x0,08 cm). The positioning of the plastic bags will cover the entire knee surface (Anterior, lateral and posterior region). After the positioning of the ice bags, they will be fixed with an elastic bandage (compression). To protect the skin against frost bites, all the knee surface will be covered with a moistened operative field (45x50x0,01 cm, 100% cotton)
  Other Names: Cold Therapy; Ice Therapy

SUMMARY:
The purpose of this case series will be to provide a detailed description of a standardized short-term cryotherapy application protocol using validated functional outcome measures in individuals with end stage KOA

DETAILED DESCRIPTION:
There are no studies determining the efficacy of cryotherapy in pain, function and quality of life for patients with end stage Knee Osteoarthritis (KOA). This case series describes a standardized treatment program for end stage patients with KOA and outcomes over a 12-week period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee osteoarthritis based on clinical and radiographic criteria of American College of Rheumatology
* Osteoarthritis signals in at least one of the compartments of the knee joint (tibiofemoral and / or the patellofemoral joint)
* Do not perform regular physical activity
* Grade 4 according to the criteria of Kellgren & Lawrence knee osteoarthritis radiographic examination scale.
* Minimum score of 4 cm in Visual Analogue Scale (total 10 cm)
* Body Mass Index less or equal to 40 kg/cm2

Exclusion Criteria:

* Physical therapy within 3 months prior to the research project
* Corticosteroid or Hyaluronic Acid injection in the knee (in the previous 6 months)
* Cardiorespiratory, neurological or other rheumatic dysfunctions associated with the diagnosis of knee osteoarthritis.
* Hip, knee or ankle surgery
* Any other type of chronic condition that can lead to pain.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (Pain scale) | Change between the baseline assessments and the Post intervention (Sixth week), 3 week follow up (9th week), 6 week follow up (12th week)
  VAS is a well recognized tool to measure the intensity of pain that visually represents the intensity of pain that the individual believes to present. The scale will be positioned in front of the individual and will have a range of 0 to 10 cm, with 0 being the complete absence of pain and 10, the maximum intensity of pain reported by the individual.

SECONDARY OUTCOMES:
Western Ontario & McMaster Universities Osteoarthritis (WOMAC) | Change between the baseline assessments and the Post intervention (Sixth week), 3 week follow up (9th week), 6 week follow up (12th week)
  WOMAC is a self-report questionnaire designed to assess the problems experienced by people with OA of the lower limb. The score for the items is expressed through a Likert scale, where the rating is calculated as: none = 0, low = 25 = 50 moderate, severe = 75 and very severe = 100. The maximum score on each section is expressed as a percentage, with higher scores indicating greater pain, stiffness and physical dysfunction. Each point corresponds to a particular dimension (pain, stiffness and physical function). This questionnaire has been translated and validated for the Portuguese language from Brazil.
40m fast paced walk test | Change between the baseline assessments and the Post intervention (Sixth week), 3 week follow up (9th week), 6 week follow up (12th week)
  Fast paced walking test that is timed by a distance of 4X10 meters, totaling 40 meters. It is used as a direct measure to correlate the ability to walk fast, short distances. Administered at a distance of 10 meters (demarcated by tapes), a cone is placed 2 meters before the start and 2 meters after the end of each marking. The participant is instructed to walk the 10 meters (from the start marking), turn around in the cone and walk another 10 meters, successively until completing the distance of 40 meters. Time is considered only between the tracks (start and end). The final score is calculated based on the speed of the participant performs the procedure and compared with normative values of healthy adults.
30-Second Chair to Stand Test | Change between the baseline assessments and the Post intervention (Sixth week), 3 week follow up (9th week), 6 week follow up (12th week)
  The 30 seconds chair stand test is administered using an armless chair, with seat height of about 43cm from the ground. The chair has a rubber for not slipping under its support and is placed against a wall to avoid oscillations. The participant sits in the middle of the chair with the back straight, feet apart, aligned with the shoulder width apart and flat on the floor at an angle slightly behind the knee line. Moreover, to help maintain balance, one foot may be slightly placed ahead of the other and arms crossed against the chest. The test consists of the greatest number of times from a sitting position to a standing over a period of 30 seconds. Thus, it is possible to evaluate a wide range of skill levels with scores ranging from 0, for those who cannot complete a single repetition and values greater than 20 reps for the well prepared individuals.
Stair climb test | Baseline assessment 1 (First week), Baseline assessment 2 (Second week), Baseline assessment 3 (Third Week), Post intervention (Sixth week), 3 week follow up (9th week), 6 week follow up (12th week)
  Test where the participant should go up and down a stair in the shortest possible time. The participant will be positioned in front of the stair, and at the therapeut sign must climb the indicated steps (12 steps), and go down, being able to use the handrail as a security instrument. The height of each stair step will be 20 cm, with a handrail, in an illuminated environment, free of traffic and external distractions. A pre-test is performed to identify the need for safety measures. The final score is calculated based on the time the participant performs the procedure and compared with the normative values available for the test
Short Form 36 | Change between the baseline assessments and the Post intervention (Sixth week), 3 week follow up (9th week), 6 week follow up (12th week)
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures.
Pain catastrophizing scale | Change between the baseline assessments and the Post intervention (Sixth week), 3 week follow up (9th week), 6 week follow up (12th week)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas O Dantas, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Federal University of São Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No